CLINICAL TRIAL: NCT07271693
Title: A Phase I, Randomized, Investigator/Participant-blind, Parallel-group, Placebo-controlled, Single and Multiple Ascending Dose Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7806881 in Healthy Participants
Brief Title: A Study to Determine the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7806881 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP46089
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RO7806881: Single Ascending Dose (SAD) (Experimental): Participants will receive single doses of RO7806881, at 8 dose levels across different cohorts.
  Interventions: Drug: RO7806881
- Placebo: SAD (Placebo Comparator): Participants will receive single doses of placebo, matched to each of the 8 dose levels of RO7806881.
  Interventions: Drug: Placebo
- RO7806881: Multiple Ascending Doses (MAD) (Experimental): Participants will receive multiple doses of RO7806881, at 4 dose levels across different cohorts, per the predefined dosing regimen.
  Interventions: Drug: RO7806881
- Placebo: MAD (Placebo Comparator): Participants will receive multiple doses of placebo, matched to each of the 4 dose levels of RO7806881, per the predefined dosing regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7806881 — RO7806881 will be administered as per the schedule specified in the protocol.
  Arms: RO7806881: Multiple Ascending Doses (MAD); RO7806881: Single Ascending Dose (SAD)
Drug: Placebo — Placebo will be administered as per the schedule specified in the protocol.
  Arms: Placebo: MAD; Placebo: SAD

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of single and multiple ascending doses of RO7806881 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or females who are overtly healthy as determined by medical evaluation
* Participants must have body weight (BW) ≥ 40 kilograms (kg) and body mass index (BMI) within the range 18-32 kilograms per square meter (kg/m^2) (inclusive)

Exclusion Criteria:

* Pregnancy, breastfeeding, or intention to become pregnant during the study or within 6 months after the final dose of study treatment
* History of any clinically significant autoimmune, gastrointestinal, renal, hepatic, pulmonary, neurological, psychiatric, cardiovascular, endocrinological, hematological, or allergic disease; metabolic disorder; cancer or cirrhosis
* Latent tuberculosis (TB) or potentially active TB
* Any major illness within 1 month before the screening examination or any febrile illness within 1 week prior to the screening visit and up to first dose administration
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study
* History of hypersensitivity to biologic agents or any of the excipients in the formulation, or other allergy that contraindicates participation in the study
* Live vaccines within 1 month of the first screening visit or during the screening period
* Non-live vaccines within 2 weeks prior to dosing
* Previous exposure to RO7806881
* Positive hepatitis C virus (HCV) antibody test result
* Positive test results for hepatitis B infection
* Positive human immunodeficiency virus (HIV) antibody test result
* Positive test result consistent with cytomegalovirus (CMV) or epstein-barr virus (EBV)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
SAD Part: Number of Participants With Adverse Events (AEs) | Up to Day 127
MAD Part: Number of Participants With AEs | Up to Day 162
SAD Part: Number of Participants With Dose-limiting Adverse Events (DLAEs) | Up to Day 127
MAD Part: Number of Participants With DLAEs | Up to Day 162

SECONDARY OUTCOMES:
SAD and MAD Parts: Serum Concentration of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Maximum Concentration (Cmax) of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Minimum Concentration (Cmin) of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Area Under the Curve (AUC) From the Last Time of Dosing to the Last Measurable Concentration (AUClast) of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Apparent Total Body Clearance (CL/F) of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Volume of Distribution at Steady-state Conditions (Vss) of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Dose Proportionality for AUC | SAD: Up to Day 127; MAD: Up to Day 162
SAD and MAD Parts: Dose Proportionality for Cmax | SAD: Up to Day 127; MAD: Up to Day 162
MAD Part: Accumulation Ratio (Racc) of RO7806881 | Up to Day 162
SAD and MAD Parts: Absolute Bioavailability of RO7806881 | SAD: Up to Day 127; MAD: Up to Day 162

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- New Zealand Clinical Research - Christchurch, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No